CLINICAL TRIAL: NCT00864175
Title: A Phase 1/2, Modified Dose Escalation, Open Label Trial to Determine the Therapeutic Effect and Safety of INCB007839 Combined With Trastuzumab in Patients With Previously Untreated HER2 Positive Metastatic Breast Cancer
Brief Title: Open Label Trial of INCB07839 to Determine Effect and Safety of INCB007839 Plus Trastuzumab in HER2 Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Incyte suspended development of the compound.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 7839-202
Record Dates: First submitted 2009-01-26; First posted 2009-03-18 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A - INCB007839 and Trastuzumab (Experimental): INCB007839 100 mg BID and trastuzumab
  In Cycle 1, trastuzumab will be administered at a loading dose of 8 mg/kg as a 90 minute intravenous infusion on Day 8. In all subsequent 21-day cycles, trastuzumab will be administered at 6 mg/kg as a 90 minute intravenous infusion on Day 1.
  Interventions: Drug: INCB007839; Drug: trastuzumab
- Treatment B - INCB007839 and Trastuzumab (Experimental): INCB007839 200 mg BID and trastuzumab
  In Cycle 1, trastuzumab will be administered at a loading dose of 8 mg/kg as a 90 minute intravenous infusion on Day 8. In all subsequent 21-day cycles, trastuzumab will be administered at 6 mg/kg as a 90 minute intravenous infusion on Day 1.
  Interventions: Drug: INCB007839; Drug: trastuzumab
- Treatment C - INCB007839 and Trastuzumab (Experimental): INCB007839 300 mg BID and trastuzumab
  In Cycle 1, trastuzumab will be administered at a loading dose of 8 mg/kg as a 90 minute intravenous infusion on Day 8. In all subsequent 21-day cycles, trastuzumab will be administered at 6 mg/kg as a 90 minute intravenous infusion on Day 1.
  Interventions: Drug: INCB007839; Drug: trastuzumab
- Treatment D - INCB007839 and Docetaxel (Experimental): INCB007839 300mg BID with docetaxel
  Interventions: Drug: INCB007839; Drug: Docetaxel

INTERVENTIONS:
Drug: INCB007839 — 100 mg BID
  Arms: Treatment A - INCB007839 and Trastuzumab
Drug: INCB007839 — 200 mg BID
  Arms: Treatment B - INCB007839 and Trastuzumab
Drug: INCB007839 — 300 mg BID
  Arms: Treatment C - INCB007839 and Trastuzumab
Drug: INCB007839 — 300 mg BID
  Arms: Treatment D - INCB007839 and Docetaxel
Drug: trastuzumab — trastuzumab will be administered at a loading dose of 8 mg/kg as a 90 minute intravenous infusion on Day 8. In all subsequent 21-day cycles, trastuzumab will be administered at 6 mg/kg as a 90 minute intravenous infusion on Day 1.
  Arms: Treatment A - INCB007839 and Trastuzumab; Treatment B - INCB007839 and Trastuzumab; Treatment C - INCB007839 and Trastuzumab
Drug: Docetaxel
  Arms: Treatment D - INCB007839 and Docetaxel

SUMMARY:
This is a single arm, modified dose escalation, open label trial with the objectives of: (1) Determining a safe optimal dose of INCB007839 in combination with trastuzumab and docetaxel (2) Determining clinical efficacy and safety of INCB007839 in combination with trastuzumab and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast carcinoma that is HER2 positive
* Measurable disease as defined by the RECIST criteria
* Life expectancy greater than or equal to 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Received any anticancer medications in the 28 days prior to enrollment into this study
* Received any anticancer medications for cancers other than breast cancer within 6 months prior to enrollment in this study.
* History of deep venous thrombosis within the last year
* Contraindication to low dose warfarin therapy
* Clinically significant cardiomyopathy
* Prior treatment with INCB007839 or trastuzumab or lapatinib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete + partial response) using RECIST (Response Evaluation Criteria in Solid Tumor) criteria | Day 1 of each completed subsequent 21-day treatment cycle and the End of Study Visit.

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetic (PK) profile of INCB007839 and trastuzumab when given in combination | Monthly
  For Cycle 1, PK samples to be collected on Day 8 and Day 15 at pre-dose the morning dose of INCB007839. For Cycles 2, 3 and 4, PK will be collected as a single sample, obtained at pre-dose, on Day 1. PK samples will not be collected at Cycle 5 or later.
  o. For Cycle 1, PD samples to be collected at time of screening and at pre-dose on Day 1, Day

CONTACTS AND LOCATIONS:
Overall Officials: Bijyoyesh Mookerjee, MD, Study Director — Incyte Corporation
Locations (12):
- India (12):
  - Visakhapatnam, Andhra Pradesh
  - New Delhi, Ansari Nagar
  - Mangalore, Attavar
  - Bangalore, Karnataka
  - Hyderabaad, Punjagutta
  - Bangalore, Ram Nagar
  - Delhi, Rohini
  - Delhi, Vasundhara Enclave
  - Bhopal
  - Kolkata
  - Nashik
  - Pune